CLINICAL TRIAL: NCT01642836
Title: Clinic, Family & Community Collaboration to Treat Overweight and Obese Children
Brief Title: Clinic, Family & Community Intervention for Children With Overweight and Obesity (Stanford GOALS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Thomas Robinson, Professor of Pediatrics and of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19311; U01HL103629 (NIH)
Record Dates: First submitted 2012-07-10; First posted 2012-07-17 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Health; Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- multi-component, multi-level, multi-setting (MMM) (Experimental): 1. a theory-based community team sports program designed specifically for overweight and obese children,
  2. a home-based family intervention to reduce screen time, alter the home food/eating environment, and promote self-regulatory skills for eating and activity behavior change, and
  3. a primary care provider behavioral counseling intervention linked to the community and home interventions.
  Interventions: Behavioral: MMM
- Health and Nutrition Education (Active Comparator): Enhanced standard care/health and nutrition education intervention:
  1. notification of primary care providers about metabolic measures and blood pressure
  2. state-of-the-art information-based health and nutrition education, including semi-annual home counseling visits, monthly health education newsletters for children and for parents/guardians, and a series of quarterly, community-based evening health lectures and "Family Fun Nights"
  Interventions: Behavioral: Health and Nutrition Education

INTERVENTIONS:
Behavioral: MMM — 1. a theory-based community team sports program designed specifically for overweight and obese children,
  2. a home-based family intervention to reduce screen time, alter the home food/eating environment, and promote self-regulatory skills for eating and activity behavior change, and
  3. a primary care provider behavioral counseling intervention linked to the community and home interventions.
  Arms: multi-component, multi-level, multi-setting (MMM)
Behavioral: Health and Nutrition Education — Enhanced standard care/health and nutrition education intervention:
  1. notification of primary care providers about metabolic measures and blood pressure
  2. state-of-the-art information-based health and nutrition education, including semi-annual home counseling visits, monthly health education newsletters for children and for parents/guardians, and a series of quarterly, community-based evening health lectures and "Family Fun Nights"
  Arms: Health and Nutrition Education

SUMMARY:
Stanford GOALS is a large-scale, community-based randomized controlled trial of an innovative, interdisciplinary, multi-component, multi-level, multi-setting (MMM) approach to treating overweight and obese children. Primary Research Question: Will a 3-year, innovative, interdisciplinary, multi-component, multi-level, multi-setting (MMM) community-based intervention to treat overweight and obese children significantly reduce BMI compared to an enhanced standard care/health and nutrition education active comparison intervention?

DETAILED DESCRIPTION:
Single-blind study with all outcomes assessors (data collectors) and Investigators masked (blinded) to intervention assignment. Intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* 7-11 years of age
* BMI greater than or equal to the 85th percentile for age and sex on the 2000 U.S. Centers for Disease Control and Prevention (CDC) BMI reference

Exclusion Criteria:

* Have been diagnosed with a medical condition affecting growth (a genetic or metabolic disease/syndrome associated with obesity, Type 1 diabetes, Type 2 diabetes taking medication, chronic gastrointestinal diseases, Chronic renal diseases, uncorrected structural heart disease, heart failure, heart transplant, anorexia nervosa or bulimia nervosa or binge eating disorder (present or past), AIDS or HIV infection, pregnancy);
* Take medications affecting growth (systemic corticosteroids more than 2 weeks in the past year, insulin, oral hypoglycemics, thyroid hormone, growth hormone);
* Have a condition limiting their participation in the interventions (e.g., unable to participate in routine physical education classes at school, requiring oxygen supplementation for exertion, developmental or physical disability preventing participation in interventions, children or parents/guardians who cannot medically participate in mild dietary restrictions and/or increased physical activity for any reason);
* Have a condition limiting participation in the assessments (child or primary caregiver not able to read surveys in English or Spanish, child two or more grade levels delayed in school for reading and writing in her native language);
* Are unable to read, understand or complete informed consent in English or Spanish;
* Plan to move from the San Francisco Bay Area within the next 36 months.
* Are deemed to have another characteristic that makes them unsuitable for participation in the study in the judgment of the Principal Investigator.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 241 (Actual)
Dates: Start 2012-07-13 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

PRIMARY OUTCOMES:
body mass index trajectory (change) | baseline, 1, 2 and 3 years
  slope of measured weight in kilograms divided by the square of height in meters

SECONDARY OUTCOMES:
waist circumference | baseline, 1, 2 and 3 years
  waist circumference in centimeters
triceps skinfold thickness | baseline, 1, 2 and 3 years
  triceps skinfold thickness in mm
Percent median BMI for age and sex (calculated from BMI) | baseline, 1, 2, and 3 years
  age- and sex-adjusted BMI
Waist-to-Height Ratio | baseline, 1, 2 and 3 years
  calculated from waist and height measures
Percent body fat (estimated) | baseline, 1, 2, and 3 years
  Estimated from regression equation
fasting Total Cholesterol, LDL-Cholesterol, HDL-Cholesterol, Triglycerides, Insulin, glucose, hemoglobin A1c, high sensitivity C-Reactive Protein, Alanine Aminotransferase (ALT) | baseline, 1, 2 and 3 years
  lab assays of fasting samples
resting blood pressure | baseline, 1, 2 and 3 years
  automated resting blood pressure
resting heart rate | baseline, 1, 2 and 3 years
  automated pulse
physical activity measured by accelerometry | baseline, 1, 2 and 3 years
  Actigraph model GT3X+ total and after school physical activity and sedentary behavior
screen time and other sedentary behaviors | baseline, 1, 2 and 3 years
  self-reported weekday, saturday and sunday, television, movies, video games, computer, portable media devices, mobile phones
Typical household Television (TV) use | baseline, 1, 2, and 3 years
  Constant TV household measure
Average total daily energy intake | baseline, 1, 2 and 3 years
  from 24 hour diet recalls
Percent of energy intake from fat | baseline, 1, 2, and 3 years
  from 24 hour diet recalls
Added sugar | baseline, 1, 2, and 3 years
  from 24 hour diet recalls
Eating with screens | baseline, 1, 2, and 3 years
  breakfast, dinner and energy (from 24-hour diet recalls)
Depressive symptoms | baseline, 1, 2 and 3 years
  Children's Depression Index short form
Weight Concerns | baseline, 1, 2 and 3 years
  Overconcern with weight and shape scale
School performance | baseline, 1, 2 and 3 years
  parent/guardian reported grades
Children's sleep habits | baseline, 1, 2 and 3 years
  parent/guardian reported
Implicit theories | baseline, 1, 2, and 3 years
  fixed versus growth mindset
Parent/guardian weight | baseline, 1, 2, and 3 years
  measured weight
Parent/guardian body mass index | baseline, 1, 2, and 3 years
  calculated from measures of height and weight
Parent/guardian waist circumference | baseline, 1, 2, and 3 years
  waist circumference measured in cm
Parent/guardian reported physical activity | baseline, 1, 2, and 3 years
  survey
Parent/guardian health literacy | baseline, 1 and 2 years
  New Vital Sign (NVS) measure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas N Robinson, MD, MPH, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators can request the limited public access data set from the National Heart, Lung, and Blood Institute Biologic Specimen and Data Repository Information Coordinating Center
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data currently available
Access Criteria: Investigators can request the limited public access data set from the National Heart, Lung, and Blood Institute Biologic Specimen and Data Repository Information Coordinating Center at https://biolincc.nhlbi.nih.gov/studies/?q=coptr
URL: https://biolincc.nhlbi.nih.gov/studies/?q=coptr

REFERENCES:
- [Background] Robinson TN, Matheson D, Desai M, Wilson DM, Weintraub DL, Haskell WL, McClain A, McClure S, Banda JA, Sanders LM, Haydel KF, Killen JD. Family, community and clinic collaboration to treat overweight and obese children: Stanford GOALS-A randomized controlled trial of a three-year, multi-component, multi-level, multi-setting intervention. Contemp Clin Trials. 2013 Nov;36(2):421-35. doi: 10.1016/j.cct.2013.09.001. Epub 2013 Sep 10. PMID 24028942
- [Derived] Robinson TN, Matheson D, Wilson DM, Weintraub DL, Banda JA, McClain A, Sanders LM, Haskell WL, Haydel KF, Kapphahn KI, Pratt C, Truesdale KP, Stevens J, Desai M. A community-based, multi-level, multi-setting, multi-component intervention to reduce weight gain among low socioeconomic status Latinx children with overweight or obesity: The Stanford GOALS randomised controlled trial. Lancet Diabetes Endocrinol. 2021 Jun;9(6):336-349. doi: 10.1016/S2213-8587(21)00084-X. Epub 2021 Apr 29. PMID 33933181
- [Derived] JaKa MM, Wood C, Veblen-Mortenson S, Moore SM, Matheson D, Stevens J, Atkins L, Michie S, Adegbite-Adeniyi C, Olayinka O, Po'e EK, Kelly AM, Nicastro H, Bangdiwala SI, Barkin SL, Pratt C, Robinson TN, Sherwood NE. Applying the Behavior Change Technique Taxonomy to Four Multicomponent Childhood Obesity Interventions. West J Nurs Res. 2021 May;43(5):468-477. doi: 10.1177/0193945920954782. Epub 2020 Sep 10. PMID 32909523
- [Derived] Truesdale KP, Matheson DM, JaKa MM, McAleer S, Sommer EC, Pratt CA. Baseline diet quality of predominantly minority children and adolescents from households characterized by low socioeconomic status in the Childhood Obesity Prevention and Treatment Research (COPTR) Consortium. BMC Nutr. 2019 Sep 9;5:38. doi: 10.1186/s40795-019-0302-y. eCollection 2019. PMID 32153951
- [Derived] Cui Z, Truesdale KP, Robinson TN, Pemberton V, French SA, Escarfuller J, Casey TL, Hotop AM, Matheson D, Pratt CA, Lotas LJ, Po'e E, Andrisin S, Ward DS. Recruitment strategies for predominantly low-income, multi-racial/ethnic children and parents to 3-year community-based intervention trials: Childhood Obesity Prevention and Treatment Research (COPTR) Consortium. Trials. 2019 May 28;20(1):296. doi: 10.1186/s13063-019-3418-0. PMID 31138278